CLINICAL TRIAL: NCT03407885
Title: The Impact of Medicare Bundled Payments: Evidence From a Nationwide Randomized Evaluation for Lower Extremity Joint Replacement
Brief Title: The Impact of Medicare Bundled Payments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Finkelstein (Other)
Collaborators: Harvard University (Other); University of Chicago (Other); Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Amy Finkelstein, Scientific Director, J-PAL North America, Abdul Latif Jameel Poverty Action Lab
Organization: Abdul Latif Jameel Poverty Action Lab (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JPAL-0740
Record Dates: First submitted 2017-10-13; First posted 2018-01-23 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Arthroplasty, Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Bundled payments for knee and hip replacement
  Interventions: Other: Bundled payments for knee and hip replacement
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Bundled payments for knee and hip replacement — The bundled payment model holds acute care hospitals (ACHs) financially responsible for the spending and quality of an entire episode of care for two types of hospital admissions: MS-DRG 469 and 470. An episode begins with an ACH stay that results in a discharge in one of the two DRGs, and ends 90 days after discharge. Before each performance year begins, hospitals receive target prices from CMS, determined by historical hospital and regional episode expenditures. Hospitals are eligible for reconciliation payment from CMS if they spend less than the target prices for an episode, provided that they met an "acceptable" quality standard. Conversely, they are responsible for paying the difference if they spend more than the target prices.
  Arms: Experimental

SUMMARY:
Bundled payments (BP) are a key part of Medicare's shift away from the traditional fee-for-service (FFS) payment model. The investigators propose to study a nationwide randomized-controlled trial (RCT) of bundled payments for knee and hip replacements that was designed and implemented by CMS and launched in April 2016. Randomization was conducted at the Metropolitan Statistical Area (MSA) level with 67 MSAs and about 800 hospitals assigned to the treatment group. The investigators will examine the impact of bundled payments on Medicare spending, utilization, and quality. Study findings should be directly relevant for the design of payments for knee and hip replacements, two common and expensive medical procedures. Average impacts, as well as variation in impact across types of providers and markets may also shed light on economic mechanisms, which should be relevant for bundled payment initiatives under consideration for other medical services.

ELIGIBILITY:
Inclusion Criteria:

* Acute care hospital paid under the inpatient prospective payment system (IPPS)
* Hospital admission for major joint replacement or reattachment of lower extremity with and without major complications or comorbidities (MS-DRG 469 and 470)

Exclusion Criteria:

* MSA exclusion criteria:
* MSAs with low volume of LEJR
* MSAs with high take-up of BPCI
* MSAs with large share of LEJR in Maryland hospitals
* Hospital exclusion criteria:
* Hospitals participating in certain models of BPCI.
* Patient exclusion criteria (the episode is cancelled if any of the following occurs during the episode):
* Patient not covered by both Medicare Parts A and B
* Patient eligibility for Medicare is due to end stage renal disease (ESRD)
* Patient is in a managed care plan
* Patient is in a United Mine Workers of America Plan
* Medicare is not the primary payer for the patient
* Patient dies during the episode
* Patient is re-admitted to an ACH for one of the two CJR DRGs during the episode
* Patient initiates an LEJR episode under BPCI during the episode
* Payments and services that occur in the episode that are excluded are:
* hemophilia clotting factors
* new technology add-on payments
* transitional pass-through payment for medical devices
* payments from certain incentive programs
* otherwise included payments that exceed two standard deviations of the regional mean
* services unrelated to the index admission as defined by CMS (including certain inpatient hospital stays, Part B services, and per beneficiary per month (PBPM) payments).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Share of LEJR admissions discharged to institutional Post-Acute Care (PAC) | At hospital discharge up to 3 days
  Share of lower extremity joint replacement (LEJR) index admissions discharged to institutional post-acute care facilities (i.e. skilled nursing facilities (SNF), long term care hospitals (LTCH) or inpatient rehabilitation facilities (IRF)). LEJR index admissions are eligible admissions at acute care hospitals (ACH) that result in a discharge in either DRG 469 or 470.

SECONDARY OUTCOMES:
Share of LEJR admissions discharged to any Post Acute Care (PAC) | At hospital discharge up to 3 days
  Share of LEJR index admissions discharged to any PAC, which includes Institutional Post Acute Care (SNF, LTCH, IRF) plus home health agency. LEJR index admissions are eligible admissions at acute care hospitals (ACH) that result in a discharge in either DRG 469 or 470.
Number of days in Institutional PAC during episode | Begins with index admission and ends 90 days post-discharge from index admission
  number of days in institutional PAC facilities (sum of length of stays in SNF, LTCH and IRF)
Total covered Medicare payments during episode | Begins with index admission and ends 90 days post-discharge from index admission
  Total covered Medicare payments are defined as the total amount of Medicare Part A and part B Fee-for-Service (FFS) payments that are included in the bundle. Note that, as defined, total covered Medicare payments are the payments that would be made in the absence of Bundled Payments (i.e. payments that would occur under FFS Medicare). These are counterfactual for the treatment MSAs. If the data become available, the investigators plan to also look at actual payments made during the episode (which would include any reconciliation payments or repayments to or from hospitals in the treatment MSAs).
Total covered Medicare payments for Institutional PAC during episode | Begins with index admission and ends 90 days post-discharge from index admission
Total covered Medicare payments for any PAC during episode | Begins with index admission and ends 90 days post-discharge from index admission
Total beneficiary payments owed out of pocket during episode | Begins with index admission and ends 90 days post-discharge from index admission

OTHER OUTCOMES:
Any THA/TKA complication | Begins with index admission and ends 90 days post-discharge from index admission
  The total hip arthroplasty/total knee arthroplasty (THA/TKA) complication measure is a facility-level risk-standardized 90-day complication rate for total hip and total knee arthroplasty and is part of the targeted quality measure. However this component of the targeted quality measure is a three-year moving average. While it may not be feasible to replicate the measure, the investigators will code the underlying the eight "complications", which are heart attack, pneumonia, or sepsis/septicemia/shock within seven days of admission, surgical site bleeding, pulmonary embolism, or death within 30 days of admission, and mechanical complications or periprosthetic joint/wound infection within 90 days of admission. The proposed measure is an indicator for whether any of the eight THA/TKA complications occur.
Number of THA/TKA complications | Begins with index admission and ends 90 days post-discharge from index admission
  The total hip arthroplasty/total knee arthroplasty (THA/TKA) complication measure is a facility-level risk-standardized 90-day complication rate for total hip and total knee arthroplasty and is part of the targeted quality measure. However this component of the targeted quality measure is a three-year moving average. While it may not be feasible to replicate the measure, the investigators will code the underlying the eight "complications", which are heart attack, pneumonia, or sepsis/septicemia/shock within seven days of admission, surgical site bleeding, pulmonary embolism, or death within 30 days of admission, and mechanical complications or periprosthetic joint/wound infection within 90 days of admission. The proposed measure is the number of THA/TKA complications that occur.
Share of LEJR admissions with an ER visit within 90-days of discharge from index admission | Begins with index admission and ends 90 days post-discharge from index admission
90-day all-cause readmission | 90 days post-discharge from index admission
Number of covered procedures | Duration of hospital stay - average 3 days
Complexity of patient mix for LEJR procedures, measured by patient demographics | Duration of hospital stay - average 3 days
  The complexity of patient mix for LEJR procedures is measured by the projected episode payment using patient demographics. The investigators will generate projected episode payment based on coefficients from a regression of episode payment on patient demographics in the pre-period, controlling for MSA fixed effect. The set of patient demographics include fully interacted five-year-age-bin, race, and sex dummies, dummy for Medicaid status, and dummy for disability.
Complexity of patient mix for LEJR procedures, measured by patient demographics and comorbidities | Duration of hospital stay - average 3 days
  The complexity of patient mix for LEJR procedures is measured by the projected episode payment using patient characteristic, including both demographic and comorbidity measures. The investigators will generate projected episode payment based on coefficients from a regression of episode payment on patient characteristics in the pre-period, controlling for MSA fixed effect. The set of patient characteristics include fully interacted five-year-age-bin, race, and sex dummies, dummy for Medicaid status, dummy for disability, dummies for Charlson comorbidities, and dummy for major complication or comorbidity (MCC).
1 year total covered Medicare payments | one year since index admission
1 year mortality | one year since index admission
1 year all-cause readmission | one year since index admission
1 year outpatient opioid use | one year since index admission

CONTACTS AND LOCATIONS:
Overall Officials: Amy N Finkelstein, PhD, Principal Investigator — Massachusetts Institute of Technology; Yunan Ji, Principal Investigator — Harvard University; Neale Mahoney, PhD, Principal Investigator — University of Chicago; Jon Skinner, PhD, Principal Investigator — Dartmouth College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finkelstein A, Ji Y, Mahoney N, Skinner J. Mandatory Medicare Bundled Payment Program for Lower Extremity Joint Replacement and Discharge to Institutional Postacute Care: Interim Analysis of the First Year of a 5-Year Randomized Trial. JAMA. 2018 Sep 4;320(9):892-900. doi: 10.1001/jama.2018.12346. PMID 30193277
- [Result] Einav L, Finkelstein A, Ji Y, Mahoney N. Randomized trial shows healthcare payment reform has equal-sized spillover effects on patients not targeted by reform. Proc Natl Acad Sci U S A. 2020 Aug 11;117(32):18939-18947. doi: 10.1073/pnas.2004759117. Epub 2020 Jul 27. PMID 32719129
- [Result] Einav L, Finkelstein A, Ji Y, Mahoney N. VOLUNTARY REGULATION: EVIDENCE FROM MEDICARE PAYMENT REFORM. Q J Econ. 2022 Feb;137(1):565-618. doi: 10.1093/qje/qjab035. Epub 2021 Sep 20. PMID 35233120